CLINICAL TRIAL: NCT04869033
Title: Effects of Farinelli's Breathing Exercise on Cardiorespiratory Fitness and Symptoms in COPD Patients
Brief Title: Effects of Farinelli's Breathing Exercise in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Wannaporn Tongtako, Ph.D., Principal investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EX PHYSIO SPSC 2
Record Dates: First submitted 2021-04-01; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: COPD Patients
Keywords: Farinelli's breathing exercise; COPD; pulmonary function; respiratory muscle strength; aerobic capacity; cytokine; COPD symptoms
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Sixteen patients with COPD (GOLD I) with mild and moderate (GOLD II) severity aged 51 - 80 years old who visited at the outpatient examination room, Phramongkutklao Hospital divided into 2 groups; diaphragmatic breathing group (DB; n=8) and Farinelli's breathing group (FB; n=8). Participants in each group were administered to complete breathing exercise 5 times per week for 8 weeks. Physiological data and pulmonary function (FVC, FEV1, PEF, FEV1/FVC, FEF25-75%, MVV, VC, TV, IRV, ERV and IC), respiratory muscle strength (MIP and MEP), aerobic capacity (6-MWD and VO2max), impact of COPD questionnaire (mMRC and CAT), cytokine (TNF-α and IL-6), and oxidative stress (MDA) were analyzed during Pre- and Post-test. The dependent variables between pre-test and post-test were analyzed by a paired t-test. Independent t-test was used to compare the variables between groups. Differences were significant at p < .05.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Farinelli's breathing group (Experimental): Complete Farinelli's breathing exercise 5 times per week for 8 weeks.
  Interventions: Other: Farinelli's Breathing Exercise
- Diaphragmatic breathing group (control group) (Other): Complete Diaphragmatic breathing exercise 5 times per week for 8 weeks.
  Interventions: Other: Diaphragmatic Breathing Exercise

INTERVENTIONS:
Other: Farinelli's Breathing Exercise — after 1 minute of normal breathing, follow this instruction; inhale 2 seconds, suspend 2 seconds, exhale 2 seconds. inhale 3 seconds, suspend 3 seconds, exhale 3 seconds. inhale 4 seconds, suspend 4 seconds, exhale 4 seconds. inhale 5 seconds, suspend 5 seconds, exhale 5 seconds. inhale 6 seconds, suspend 6 seconds, exhale 6 seconds. This cycle lasted 1 minute (60 seconds), called Farinelli's breathing (FB). When participants finished these cycle, repeated it again 4 times. 1 minute of NB + 4 minutes of FB called 1 set. The participants were asked to practice 6 sets/day, 5 days/week (Monday-Friday) for week 1-4, and increased duration to 8 sets/day, 5 days/week for week 5-8.
  Arms: Farinelli's breathing group
Other: Diaphragmatic Breathing Exercise — after 1 minute of normal breathing, inhale 2 seconds and exhale 2 seconds with nasal airway. Continued breathing this pattern until 4 minutes, then back to normal breathing 1 minute . 1 minute of NB + 4 minute of DB called 1 set. The participants were asked to practice 6 sets/day, 5 days/week (Monday-Friday) for week 1-4, and increased duration to 8 sets/day, 5 days/week for week 5-8.
  Arms: Diaphragmatic breathing group (control group)

SUMMARY:
This study was to investigate the effect of Farinelli's breathing exercise on pulmonary function, respiratory muscle strength, aerobic capacity, impact of COPD questionnaires, cytokines, and oxidative stress in patients with Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Sixteen patients with COPD (GOLD I) with mild and moderate (GOLD II) severity aged 51 - 80 years old who visited at the outpatient examination room, Phramongkutklao Hospital divided into 2 groups; diaphragmatic breathing group (DB; n=8) and Farinelli's breathing group (FB; n=8). Participants in each group were administered to complete breathing exercise 5 times per week for 8 weeks. Physiological data and pulmonary function (FVC, FEV1, PEF, FEV1/FVC, FEF25-75%, MVV, VC, TV, IRV, ERV and IC), respiratory muscle strength (MIP and MEP), aerobic capacity (6-MWD and VO2max), impact of COPD questionnaire (mMRC and CAT), cytokine (TNF-α and IL-6), and oxidative stress (MDA) were analyzed during Pre- and Post-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients with COPD who treated in Phramongkutklao Hospital
* Have a history of smoking
* FEV1 predicted after bronchodilator more than 50%
* No change in medication in 4 weeks
* No history of acute exacerbation in 4 weeks
* No history of cardiac disease.

Exclusion Criteria:

* Recurrent of acute exacerbation
* Cannot participate at least 80% of training program (≤ 32 sessions of 40 sessions)
* Unwilling to continue practicing.

Ages: 51 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Force Vital Capacity (FVC) change | Change from Baseline Force Vital Capacity at 8 weeks.
  FVC is the total volume of air that can be exhaled during a maximal forced expiration effort. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FVC is measured in liters.
Forced expiratory volume in 1 second (FEV1) change | Change from Baseline Forced expiratory volume in 1 second at 8 weeks.
  FEV1 is the volume of air exhaled in the first second under force after a maximal inhalation. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEV1 was showed in liters.
Tidal Volume (TV) change | Change from Baseline Tidal Volume at 8 weeks.
  TV is the volume of air inhaled or exhaled during each respiratory cycle. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. TV is measured in liters.
Inspiratory Reserve Volume (IRV) change | Change from Baseline Inspiratory Reserve Volume at 8 weeks.
  IRV is the maximal volume of air inhaled from end-inspiration. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. IRV is measured in liters.
Expiratory Reserve Volume (ERV) change | Change from Baseline Expiratory Reserve Volume at 8 weeks.
  ERV is the maximal volume of air exhaled from end-expiration. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. ERV is measured in liters.
Inspiratory capacity (IC) change | Change from Baseline Inspiratory Capacity at 8 weeks.
  IC is the amount of air that can be inhaled after the end of a normal expiration. It is, therefore, the sum of the tidal volume and inspiratory reserve volume. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. IC was showed in liters.
Peak Expiratory Flow (PEF) change | Change from Baseline Peak Expiratory Flow at 8 weeks.
  PEF is the amount and rate of air that can be forcefully breathed out of the lungs. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. PEF is measured in liters/seconds.
Forced Expiratory Flow from 25% to 75% of vital capacity (FEF25-75%) change | Change from Baseline Forced Expiratory Flow from 25% to 75% of vital capacity (FEF25-75%) at 8 weeks.
  FEF25-75% is the average flow from the point at which 25 percent of the FVC has been exhaled to the point at which 75 percent of the FVC has been exhaled. The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEF25-75% is measured in liters/seconds.
The ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) change | Change from Baseline The ratio of forced expiratory volume in 1 second to forced vital capacity at 8 weeks.
  It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC). The participants were asked to wear a nose clip while sitting on a chair, and the researcher gave the participants the step-by-step protocol to prevent an incorrect maneuver. For the FVC maneuver, three cycles of slow normal breathing were performed before demonstrating forced inspiration and expiration. FEV1/FVC was showed in percentage.
Respiratory muscle strength change | Change from Baseline respiratory muscle strength at 8 weeks.
  Respiratory muscle strength was assessed by measuring Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP) in cmH2O. The participants were in a sitting position using a portable handheld mouth pressure meter (i.e., MicroRPM) with a nose clip. For the MIP measurement, the participants were asked to exhale until they felt no air remaining in their lungs (starting with the functional residual capacity [FRC] point), then held the device on their mouth and inhaled forcefully for 1-2 seconds. For the MEP measurement, the participants were asked to inhale until their lungs were completely filled with air (starting with the total lung capacity [TLC] point), then they kept the device on their mouth and exhaled forcefully for 1-2 seconds
Maximal Voluntary Ventilation (MVV) change | Change from Baseline Maximum Voluntary Ventilation at 8 weeks.
  The participants were asked to inhale and exhale quickly and forcefully for 10 seconds. Maximal Voluntary Ventilation (MVV) were measured in liters/minutes.
Impact of COPD change | Change from Baseline Impact of COPD at 8 weeks.
  The impact of COPD was assessed using the mMRC and the CAT. The mMRC has a 5-point (0-4) scale based on the severity of dyspnea, whereas the CAT is a patient-completed instrument to assess and quantify the quality of life and burden of the symptoms in patients with COPD. It consists of eight questions, each of which had a semantic 6-point (0-5) differential scale, providing a total score of up to 40 points. The scores 0-10, 11-20, 21-30, and 31-40 represented mild, moderate, severe, and very severe clinical impact, respectively.

SECONDARY OUTCOMES:
Cytokines change | Change from baseline cytokines at 8 weeks.
  The participants were asked for intravenous blood puncture 5 cc. The levels of cytokines (Tumor necrosis factor alpha;TNF-α and Interluekin-6; IL-6 were measured in pg/ml) were determined by using the multiplex inflammation from the plasma.
Malondialdehydes (MDA) change | Change from baseline Malondialdehydes at 8 weeks.
  The participants were asked for intravenous blood puncture 5 cc. Malondialdehydes (MDA) was analyzed by the lipid peroxidation (MDA) fluorometric assay kit in μmol/L.
Aerobic capacity change | Change from Baseline aerobic capacity at 8 weeks.
  Aerobic capacity was assessed using the 6-MWD, following the guidelines of the 2002 ATS. A modified settlement of the 25 m straight walking test with turning points. Participants were asked to wear comfortable clothes and shoes during the test, and their vital signs (i.e., resting heart rate and blood pressure) were evaluated before and after the test. The participants were asked to walk at a comfortable pace for 6 minutes under the supervision of a nurse and were permitted to terminate and rest during the test if they sensed heavy dyspnea.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Sports Science, Chulalongkorn University, Bangkok, Thailand

REFERENCES:
- [Background] Barnes PJ. Inflammatory mechanisms in patients with chronic obstructive pulmonary disease. J Allergy Clin Immunol. 2016 Jul;138(1):16-27. doi: 10.1016/j.jaci.2016.05.011. Epub 2016 May 27. PMID 27373322
- [Background] Beavers KM, Brinkley TE, Nicklas BJ. Effect of exercise training on chronic inflammation. Clin Chim Acta. 2010 Jun 3;411(11-12):785-93. doi: 10.1016/j.cca.2010.02.069. Epub 2010 Feb 25. PMID 20188719
- [Background] Cahalin LP, Braga M, Matsuo Y, Hernandez ED. Efficacy of diaphragmatic breathing in persons with chronic obstructive pulmonary disease: a review of the literature. J Cardiopulm Rehabil. 2002 Jan-Feb;22(1):7-21. doi: 10.1097/00008483-200201000-00002. PMID 11839992
- [Background] Gosselink R. Breathing techniques in patients with chronic obstructive pulmonary disease (COPD). Chron Respir Dis. 2004;1(3):163-72. doi: 10.1191/1479972304cd020rs. PMID 16281658
- [Background] Holland AE, Hill CJ, Jones AY, McDonald CF. Breathing exercises for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD008250. doi: 10.1002/14651858.CD008250.pub2. PMID 23076942
- [Background] Ksinopoulou H, Hatzoglou C, Daniil Z, Gourgoulianis K, Karetsi H. Respiratory function in vocal soloists, opera singers and wind instrument musicians. Med Lav. 2016 Dec 13;107(6):437-443. PMID 27976662
- [Background] Leelarungrayub J, Puntumetakul R, Sriboonreung T, Pothasak Y, Klaphajone J. Preliminary study: comparative effects of lung volume therapy between slow and fast deep-breathing techniques on pulmonary function, respiratory muscle strength, oxidative stress, cytokines, 6-minute walking distance, and quality of life in persons with COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 5;13:3909-3921. doi: 10.2147/COPD.S181428. eCollection 2018. PMID 30584292